CLINICAL TRIAL: NCT00094965
Title: Phase II Trial of Oxaliplatin in Combination With Bolus/Infusional 5FU/LV (FOLFOX4) in Patients With Advanced Gastrointestinal (GI) Cancers With Varying Degrees of Renal Impairment
Brief Title: Oxaliplatin With FOLFOX4 in Patients With Normal and Abnormal Renal Function
Acronym: FOLFOX4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POP5347
Record Dates: First submitted 2004-10-28; First posted 2004-10-29 (Estimated); Last update posted 2009-03-30 (Estimated); Status verified 2009-03

CONDITIONS: Gastrointestinal Cancer
Keywords: Advanced Gastrointestinal tumors and normal to severely abnormal renal function
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Oxaliplatin

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Oxaliplatin (SR96669)

INTERVENTIONS:
Drug: Oxaliplatin (SR96669) — oxaliplatin in combination with FOLFOX4

SUMMARY:
This trial is a phase II study in patients with advanced gastrointestinal (GI) malignancies who will be assigned to one of 4 cohorts (normal, mild, moderate and several renal dysfunction) based on their baseline measured creatinine clearance then treated with FOLFOX4.

Standard bone marrow and liver function inclusion and exclusion criteria must be met prior to study treatment. FOLFOX4 in the study is given every 2 weeks (1 cycle = 2 weeks) for up to 12 cycles unless there are treatment delays to allow for recovery from toxic effects. Dose modifications are included for protocol specified toxicities. After 12 treatment cycles on study, patients who are having a beneficial disease response may continue to have oxaliplatin supplied off study to continue the treatment regimen until disease progression, prohibitive toxicity or death.

Oxaliplatin pharmacokinetic studies (plasma and urine) are planned during cycles 1 and 2 on each patient. Creatinine clearance will be assessed every 2 cycles and disease status will be assessed every 3 cycles of treatment during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed locally advanced or metastatic gastrointestinal (GI) malignancy;
* Patients may have measurable or non-measurable disease;
* Prior chemotherapy, radiation therapy, hormonal therapy and immunotherapy are allowed, with the exception that patients cannot have had prior treatment with oxaliplatin, cisplatin or other nephrotoxic anticancer agent;
* Patients must have had no chemotherapy or radiotherapy within 4 weeks (28 days) prior to entering the study;
* Age 18 or older;
* Karnofsky performance status of 70% or greater for patients with normal or mildly abnormal renal function and 50% or greater for patients with moderately or severely abnormal renal function;
* Life expectancy of at least 3 months;
* Adequate bone marrow function (WBC > or = 3000 cells/mm3, ANC > or = 1500 cells/mm3, platelets > or = 100,000 cells/mm3);
* Adequate liver function (total bilirubin < or =1.5 times the institutional upper limit of normal (IULN), AST (SGOT)/ALT (SGPT) < or = 2 times the IULN, unless liver metastases are present and documented at baseline by CT or MRI scan (< or = 5 times IULN in that case), alkaline phosphatase < or = 2 times the IULN, unless liver metastases are present and documented at baseline by CT or MRI scan (< or = 5 times IULN in that case));
* Patients may have a Grade 1 neurotoxicity at study entry. Absence of deep tendon reflexes as a sole neurological abnormality does not render the patient ineligible;
* If female, not pregnant or lactating at inclusion. Documentation of a negative serum HCG pregnancy test for women of child bearing potential is required at inclusion;
* Women of child bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry, for the duration of study participation and for 6 months after discontinuation of study treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately;
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with active hydronephrosis (patients with a functioning ureteral stent are allowed on study);
* Patients who have had chemotherapy or radiotherapy within 4 weeks (28 days) prior to entering the study;
* Patients who have had a major surgery within 4 weeks (28 days) prior to entering the study;
* Patients who had prior therapy with oxaliplatin, cisplatin or other nephrotoxic anticancer agent;
* History of allergy to platinum compounds;
* Patients undergoing therapy with other investigational agents. Patients who received any investigational drug must have discontinued the investigational drug 30 days or more before beginning treatment on this study;
* Patients with known dihydropyrimidine dehydrogenase (DPD) deficiency;
* Patients who have had a history of cardiac toxicities while on 5FU/LV therapy or myocardial infarction < or = 6 months prior to study entry;
* Patients with known brain metastases because of their poor prognosis and because they often develop progressive neurological dysfunction that would confound the evaluation of neurological and other toxicities;
* Patients with interstitial pneumonia or extensive and symptomatic fibrosis of the lungs;
* Patients with uncontrolled intercurrent illness (high blood pressure, unstable angina pectoris, symptomatic congestive heart failure (NYHA III or IV), severe cardiac arrhythmia, uncontrolled diabetes or active infection);
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Adverse events. | 12 Cycles

SECONDARY OUTCOMES:
Pharmacokinetics. | 2 Cycles
Tumor evaluations for response or progressive disease. | 12 Cycles

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States